CLINICAL TRIAL: NCT00311116
Title: Serial Controlled N-of-1 Trials of Topical Vitamin E as Prophylaxis for Chemotherapy-induced Oral Mucositis in Pediatric Patients
Brief Title: Vitamin E to Prevent Mucositis in Children With Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian Feldman, Division Head, Rheumatology, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 0020010130
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Cancer
Keywords: Vitamin E; Cancer; pediatrics; supportive care; oral mucositis; Bayesian analysis; N-of-1 trial; prophylaxis
MeSH Terms: conditions — Neoplasms; Stomatitis | interventions — Vitamin E

INTERVENTIONS:
Drug: Vitamin E

SUMMARY:
The primary objective is to determine whether in children undergoing doxorubicin-containing chemotherapy, if topical vitamin E, when compared to placebo, decreases an objective measurement of oral mucositis.

DETAILED DESCRIPTION:
Oral mucositis is a common consequence of chemotherapy and is an important sequela of cancer therapy because it is painful and affects quality of life, may lead to hospitalization for hydration or pain control, and provides a portal of entry for oral microflora. In addition, oral mucositis has become a major dose-limiting toxicity and consequently, may limit delivery of anti-cancer therapy.

Despite the frequency of mucositis, there are no feasible therapies proven to be successful in preventing mucositis in children. Vitamin E is a fat-soluble essential vitamin that may protect against doxorubicin-induced oral mucositis through its anti-oxidant properties.

In this study, we will examine the efficacy of topical vitamin E as prophylaxis against chemotherapy-induced mucositis with a novel methodology appropriate for the study of rare conditions, namely combining N-of-1 trials using Bayesian meta-analysis.

The primary outcome is an objective mucositis score measured on days 7, 10, 14 and 17. Secondary outcomes included daily pain and swallowing visual analogue scale scores, and World Health Organization mucositis scores collected on days 5 to 20.

Comparisons: Objective and subjective mucositis scores will be compared in cycles associated with topical vitamin E versus cycles associated with placebo administration. We will use repeated measures analysis within a Bayesian framework in order to conduct this comparison.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cancer and treated at the Hospital for Sick Children, Toronto, Canada
* planned chemotherapy includes at least two identical courses of doxorubicin-containing chemotherapy in which the dose of doxorubicin was at least 60 mg/m2 per course
* at least 6 years of age and less than 18 years
* lives in the Greater Toronto area

Exclusion Criteria:

* allergy to vitamin E or placebo ingredients
* child is unable to comply with topical vitamin E application
* cild is receiving head or neck irradiation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16
Dates: Start 2002-07; Study Completion 2005-02

PRIMARY OUTCOMES:
Objective mucositis score at 7, 10, 14, and 17 days post initiation of chemotherapy

SECONDARY OUTCOMES:
Pain visual analogue scale
Difficulty swallowing visual analogue scale
World Health Organization mucositis grade
Analgesia use (topical, systemic non-narcotic or narcotic
Receipt of intravenous fluid, and total parenteral nutrition.
Chemotherapy decrements or delays due to mucositis

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Feldman, MD, MSc, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada